CLINICAL TRIAL: NCT06795945
Title: Evaluate the Safety of a Bovine Thymus Nuclear Extract
Brief Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel Study to Evaluate the Safety of a Bovine Thymus Nuclear Extract
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Standard Process Inc. (Industry)
Collaborators: Nutrasource Pharmaceutical and Nutraceutical Services, Inc. (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: S01-24-01-T0071
Record Dates: First submitted 2025-01-06; First posted 2025-01-28 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Immunology
Keywords: Bovine Thymus Nuclear Extract; Safety; Tolerability; Immune health

STUDY DESIGN:
Intervention Model Description: The study includes four groups: three test product groups and one placebo group (PL), all consisting of healthy male and female adults aged 18 to 65 (inclusive). Each participant's involvement in the study will last up to 25 weeks.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- TPG1 (Active Comparator): Thymus Nuclear Extract Dose 1
  Interventions: Dietary Supplement: TPG1
- TPG2 (Active Comparator): Thymus Nuclear Extract Dose 2
  Interventions: Dietary Supplement: TPG2
- TPG3 (Active Comparator): Thymus Nuclear Extract Dose 3
  Interventions: Dietary Supplement: TPG3
- PL (Placebo Comparator): Placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: TPG1 — * Thymus Nuclear Extract Dose 1 (860 mg [2 tablets, 2x/day; total 4 tablets per day])
  * Placebo (6 tablets, 2x/day; total 12 tablets per day)
  Arms: TPG1
Dietary Supplement: TPG2 — * Thymus Nuclear Extract Dose 2 (2150 mg [5 tablets, 2x/day; total 10 tablets per day])
  * Placebo (3 tablets, 2x/day; total 6 tablets per day)
  Arms: TPG2
Dietary Supplement: TPG3 — Thymus Nuclear Extract Dose 3 (3440 mg [8 tablets, 2x/day; total 16 tablets per day])
  Arms: TPG3
Dietary Supplement: Placebo — Placebo (8 tablets, 2x/day; total 16 tablets per day)
  Arms: PL

SUMMARY:
The goal of this trial is to find out if Thymus Nuclear Extract is safe and well-tolerated in healthy men and women by testing three different dose levels and comparing the results to a placebo.

DETAILED DESCRIPTION:
This is a 12 to 25 week study (if study participants are willing to follow up on study results) where participants are randomly assigned to groups and neither they nor the researchers know who receives Thymus Nuclear Extract or a placebo. The trial focuses on evaluating the safety of the extract in healthy adults by monitoring for adverse events and conducting safety assessments throughout the study.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female participants who are between 18 - 65 years of age (inclusive).
2. In good general health (i.e., no uncontrolled diseases or conditions) as deemed by the investigator and are able to consume the study product.
3. Have a body mass index (BMI) range of 18.5 - 29.9 kg/m2 (inclusive).
4. Agree to follow the restrictions on concomitant treatments as listed.
5. Agree to use acceptable contraceptive methods as listed.
6. Willing and able to agree to the requirements of this study, be willing to give voluntary consent, be able to understand and read the questionnaires, and carry out all study-related procedures.
7. Agree to the dosage instructions including the oral consumption of 8 tablets twice daily.

Exclusion Criteria:

1. Individuals who are lactating, pregnant or planning to become pregnant during the study, or demonstrates a positive pregnancy test at Visit 2.
2. Have a known sensitivity, intolerability, or allergy (especially to bovine products) to any of the study products or their excipients.
3. Have Type I diabetes, uncontrolled Type II diabetes, uncontrolled high blood pressure (≥140 systolic or ≥90 diastolic mmHg), or uncontrolled thyroid disease ("uncontrolled" defined as being unmedicated, have an unstable use of medication within 3 months prior to screening, or have a stable use of medication for 3 months but still have uncontrolled conditions).
4. Have a chronic inflammatory condition (e.g., rheumatoid arthritis, lupus, or multiple-sclerosis).
5. Have a neurological disorder which may impact cognitive testing (e.g., traumatic brain injury, epilepsy, neurodegenerative diseases).
6. Have received an organ transplant or other forms of allografts or xenografts.
7. Participants with sleep disorders (e.g., insomnia, sleep apnea, restless legs syndrome, narcolepsy, or any other condition that significantly affects sleep quality and duration)
8. Have medical condition(s) known to interfere with absorption, distribution, metabolism, or excretion of the study product (e.g., Crohn's disease, short bowel, acute or chronic pancreatitis, or pancreatic insufficiency).
9. Have a history of heart/cardiovascular disease, renal disease (dialysis or renal failure), hepatic impairment/disease, immune disorders and/or immunocompromised (i.e., HIV/AIDS).
10. Have a history of cancer (except localized skin cancer without metastases or in situ cervical cancer), unless recovery occurred more than 5 years before the screening visit.
11. Are receiving treatments for or have been hospitalized in the last 12 months for psychiatric disorders (e.g., depression, bipolar disorder, schizophrenia, etc.).
12. Reports a clinically significant illness during the 28 days before the first dose of study product.
13. Major surgery in 3 months prior to screening or planned major surgery during the study.
14. Have a history of alcohol or substance abuse in the 12 months prior to screening (including having been hospitalized for such in an in-patient or out-patient intervention program) or use that in the opinion of the investigator may be of a concern for the study.
15. Current enrollment or past participation in another study with any product(s) with at least one active ingredient within 28 days before first dose of study product or longer, if the previous test product is deemed by the investigator to have lasting effects that might influence the eligibility criteria or outcomes of current study.
16. Any other medical condition/situation or use of medications/supplements/therapies that, in the opinion of the investigator, may adversely affect the participant's ability to participate in the study or its measures or pose a significant risk to the participant.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2025-02-04 (Actual); Primary Completion 2025-11-24 (Actual); Study Completion 2025-11-24 (Actual)

PRIMARY OUTCOMES:
To assess the safety and tolerability of Thymus Nuclear Extract at 3 dose levels | 12 weeks
  Heart rate (bpm)
To assess the safety and tolerability of Thymus Nuclear Extract at 3 dose levels | 12 weeks
  Blood pressure (mmHg)
To assess the safety and tolerability of Thymus Nuclear Extract at 3 dose levels | 12 weeks
  Weight (kg)
To assess the safety and tolerability of Thymus Nuclear Extract at 3 dose levels | 12 weeks
  Body mass index (kg/m2)
To assess the safety and tolerability of Thymus Nuclear Extract at 3 dose levels. | 12 weeks
  Whole blood hemoglobin (g/dL)
To assess the safety and tolerability of Thymus Nuclear Extract at 3 dose levels | 12 weeks
  Hematocrit (%)
To assess the safety and tolerability of Thymus Nuclear Extract at 3 dose levels | 12 weeks
  Red Blood Cell Count
To assess the safety and tolerability of Thymus Nuclear Extract at 3 dose levels | 12 weeks
  Red Cell Distribution Width
To assess the safety and tolerability of Thymus Nuclear Extract at 3 dose levels | 12 weeks
  Mean Corpuscular Volume
To assess the safety and tolerability of Thymus Nuclear Extract at 3 dose levels | 12 weeks
  Mean Corpuscular Hemoglobin
To assess the safety and tolerability of Thymus Nuclear Extract at 3 dose levels | 12 weeks
  Mean Corpuscular Hemoglobin Concentration
To assess the safety and tolerability of Thymus Nuclear Extract at 3 dose levels | 12 weeks
  White Blood Cell Count and Differential
To assess the safety and tolerability of Thymus Nuclear Extract at 3 dose levels | 12 weeks
  Platelet Count
To assess the safety and tolerability of Thymus Nuclear Extract at 3 dose levels | 12 weeks
  Mean Platelet Volume
To assess the safety and tolerability of Thymus Nuclear Extract at 3 dose levels | 12 weeks
  Blood Urea Nitrogen
To assess the safety and tolerability of Thymus Nuclear Extract at 3 dose levels | 12 weeks
  Creatinine
To assess the safety and tolerability of Thymus Nuclear Extract at 3 dose levels | 12 weeks
  Estimated Glomerular Filtration rate
To assess the safety and tolerability of Thymus Nuclear Extract at 3 dose levels | 12 weeks
  Alkaline Phosphatase
To assess the safety and tolerability of Thymus Nuclear Extract at 3 dose levels | 12 weeks
  Bilirubin Total
To assess the safety and tolerability of Thymus Nuclear Extract at 3 dose levels | 12 weeks
  Aspartate Aminotransferase
To assess the safety and tolerability of Thymus Nuclear Extract at 3 dose levels | 12 weeks
  Alanine Aminotransferase
To assess the safety and tolerability of Thymus Nuclear Extract at 3 dose levels | 12 weeks
  Albumin
To assess the safety and tolerability of Thymus Nuclear Extract at 3 dose levels | 12 weeks
  Total Protein
To assess the safety and tolerability of Thymus Nuclear Extract at 3 dose levels | 12 weeks
  Globulin
To assess the safety and tolerability of Thymus Nuclear Extract at 3 dose levels | 12 weeks
  Fasting Glucose Serum
To assess the safety and tolerability of Thymus Nuclear Extract at 3 dose levels | 12 weeks
  Chloride
To assess the safety and tolerability of Thymus Nuclear Extract at 3 dose levels | 12 weeks
  Sodium
To assess the safety and tolerability of Thymus Nuclear Extract at 3 dose levels | 12 weeks
  Potassium
To assess the safety and tolerability of Thymus Nuclear Extract at 3 dose levels | 12 weeks
  Reports of adverse events

OTHER OUTCOMES:
To assess the impact of Thymus Nuclear Extract at 3 dose levels on general health (sleep and cognition) | 12 weeks
  PROMIS Disturbance - short Form 8b score
To assess the impact of Thymus Nuclear extract at 3 dosage levels on transcriptome | 25 weeks
  Whole Blood Transcriptome Analysis
To assess the impact of Thymus Nuclear Extract at 3 dose levels on general health (sleep and cognition) | 12 weeks
  Patient Health Questionnaire (PHQ-9) score
To assess the impact of Thymus Nuclear Extract at 3 dose levels on general health (sleep and cognition) | 12 weeks
  Self-Administered Gerocognitive Examination (SAGE) score
To assess the impact of Thymus Nuclear Extract at 3 dose levels on blood biomarkers | 25 weeks
  Adrenal hormones:dehydroepiandrosterone
To assess the impact of Thymus Nuclear Extract at 3 dose levels on blood biomarkers | 25 weeks
  Estradiol
To assess the impact of Thymus Nuclear Extract at 3 dose levels on blood biomarkers | 25 weeks
  Sex Hormone-Binding Globulin
To assess the impact of Thymus Nuclear Extract at 3 dose levels on blood biomarkers | 25 weeks
  Spermidine
To assess the impact of Thymus Nuclear Extract at 3 dose levels on blood biomarkers | 25 weeks
  Spermine
To assess the impact of Thymus Nuclear Extract at 3 dose levels on blood biomarkers | 25 weeks
  Putrescine
To assess the impact of Thymus Nuclear Extract at 3 dose levels on blood biomarkers | 25 weeks
  Histamine
To assess the impact of Thymus Nuclear Extract at 3 dose levels on blood biomarkers | 25 weeks
  Serotonin
To assess the impact of Thymus Nuclear Extract at 3 dose levels on blood biomarkers | 25 weeks
  Tryptamine
To assess the impact of Thymus Nuclear Extract at 3 dose levels on blood biomarkers | 25 weeks
  Tyramine
To assess the impact of Thymus Nuclear Extract at 3 dose levels on blood biomarkers | 25 weeks
  Cadaverine
To assess the impact of Thymus Nuclear Extract at 3 dose levels on blood biomarkers | 25 weeks
  Ferritin
To assess the impact of Thymus Nuclear Extract at 3 dose levels on blood biomarkers | 25 weeks
  Phosphorus
To assess the impact of Thymus Nuclear Extract at 3 dose levels on blood biomarkers | 25 weeks
  Calcium
To assess the impact of Thymus Nuclear Extract at 3 dose levels on blood biomarkers | 25 weeks
  Magnesium
To assess the impact of Thymus Nuclear Extract at 3 dose levels on blood biomarkers | 25 weeks
  Vitamin D
To assess the impact of Thymus Nuclear Extract at 3 dose levels on blood biomarkers | 25 weeks
  Vitamin B12
To assess the impact of Thymus Nuclear Extract at 3 dose levels on blood biomarkers | 25 weeks
  Folate
To assess the impact of Thymus Nuclear Extract at 3 dose levels on blood biomarkers | 25 weeks
  Homocysteine
To assess the impact of Thymus Nuclear Extract at 3 dose levels on blood biomarkers | 25 weeks
  IgM
To assess the impact of Thymus Nuclear Extract at 3 dose levels on blood biomarkers | 25 weeks
  IgA
To assess the impact of Thymus Nuclear Extract at 3 dose levels on blood biomarkers | 25 weeks
  IgG
To assess the impact of Thymus Nuclear Extract at 3 dose levels on blood biomarkers | 25 weeks
  Rheumatoid Factor
To assess the impact of Thymus Nuclear Extract at 3 dose levels on blood biomarkers | 25 weeks
  Anti-Citrullinated Protein Antibodies
To assess the impact of Thymus Nuclear Extract at 3 dose levels on blood biomarkers | 25 weeks
  Induction of Autoantibodies Against Citrullinated and Non-Citrullinated Collagen
To assess the impact of Thymus Nuclear Extract at 3 dose levels on blood biomarkers | 25 weeks
  Induction of Autoantibodies Against Citrullinated and Con-Citrullinated Fibronectin
To assess the impact of Thymus Nuclear Extract at 3 dose levels on blood biomarkers | 25 weeks
  Induction of Autoantibodies Against Citrullinated and Non-Citrullinated Vimentin
To assess the impact of Thymus Nuclear Extract at 3 dose levels on blood biomarkers | 25 weeks
  Induction of Autoantibodies Against Citrullinated and Non-Citrullinated GFAP
To assess the impact of Thymus Nuclear Extract at 3 dose levels on blood biomarkers | 25 weeks
  Induction of Autoantibodies Against Citrullinated and Non-Citrullinated Myelin Basic Protein
To assess the impact of Thymus Nuclear Extract at 3 dose levels on blood biomarkers | 25 weeks
  Induction of Autoantibodies Against Citrullinated and Non-Citrullinated Neuron-Specific Enolase
To assess the impact of Thymus Nuclear Extract at 3 dose levels on blood biomarkers | 25 weeks
  Induction of Autoantibodies Against Citrullinated and Non-Citrullinated S100 Calcium-Binding Protein B
To assess the impact of Thymus Nuclear Extract at 3 dose levels on blood biomarkers | 25 weeks
  Induction of Autoantibodies Against Citrullinated and Non-Citrullinated Intracellular Adhesion Molecule
To assess the impact of Thymus Nuclear Extract at 3 dose levels on blood biomarkers | 25 weeks
  Induction of Autoantibodies Against Citrullinated and Non-Citrullinated Brain-Derived Neurotrophic Factor
To assess the impact of Thymus Nuclear Extract at 3 dose levels on blood biomarkers | 25 weeks
  Induction of Autoantibodies Against Citrullinated and Non-Citrullinated Actin
To assess the impact of Thymus Nuclear Extract at 3 dose levels on blood biomarkers | 25 weeks
  Induction of Autoantibodies Against Citrullinated and Non-Citrullinated Zonulin
To assess the impact of Thymus Nuclear Extract at 3 dose levels on blood biomarkers | 25 weeks
  Induction of Autoantibodies Against Citrullinated and Non-Citrullinated Myosin Heavy Chain 7
To assess the impact of Thymus Nuclear Extract at 3 dose levels on blood biomarkers | 25 weeks
  Induction of Autoantibodies Against Citrullinated and Non-Citrullinated Myoglobin
To assess the impact of Thymus Nuclear Extract at 3 dose levels on blood biomarkers | 25 weeks
  Induction of Autoantibodies Against Citrullinated and Non-Citrullinated Troponin
To assess the impact of Thymus Nuclear Extract at 3 dose levels on blood biomarkers | 25 weeks
  Triglycerides
To assess the impact of Thymus Nuclear Extract at 3 dose levels on blood biomarkers | 25 weeks
  Total Cholesterol
To assess the impact of Thymus Nuclear Extract at 3 dose levels on blood biomarkers | 25 weeks
  Low-Density Lipoprotein Cholesterol
To assess the impact of Thymus Nuclear Extract at 3 dose levels on blood biomarkers | 25 weeks
  High-Density Lipoprotein Cholesterol
To assess the impact of Thymus Nuclear Extract at 3 dose levels on blood biomarkers | 25 weeks
  Apolipoprotein A
To assess the impact of Thymus Nuclear Extract at 3 dose levels on blood biomarkers | 25 weeks
  Lipoprotein A
To assess the impact of Thymus Nuclear Extract at 3 dose levels on blood biomarkers | 25 weeks
  Apolipoprotein B
To assess the impact of Thymus Nuclear Extract at 3 dose levels on blood biomarkers | 25 weeks
  IL-1
To assess the impact of Thymus Nuclear Extract at 3 dose levels on blood biomarkers | 25 weeks
  IL-1 receptor antagonist protein (IL-1RN)
To assess the impact of Thymus Nuclear Extract at 3 dose levels on blood biomarkers | 25 weeks
  IL-6
To assess the impact of Thymus Nuclear Extract at 3 dose levels on blood biomarkers | 25 weeks
  IL-8
To assess the impact of Thymus Nuclear Extract at 3 dose levels on blood biomarkers | 25 weeks
  IL-13
To assess the impact of Thymus Nuclear Extract at 3 dose levels on blood biomarkers | 25 weeks
  IL-18
To assess the impact of Thymus Nuclear Extract at 3 dose levels on blood biomarkers | 25 weeks
  IFN-alpha
To assess the impact of Thymus Nuclear Extract at 3 dose levels on blood biomarkers | 25 weeks
  IFN-beta
To assess the impact of Thymus Nuclear Extract at 3 dose levels on blood biomarkers | 25 weeks
  TGF-beta
To assess the impact of Thymus Nuclear Extract at 3 dose levels on blood biomarkers | 25 weeks
  TNF
To assess the impact of Thymus Nuclear Extract at 3 dose levels on blood biomarkers | 25 weeks
  Serum Amyloid A
To assess the impact of Thymus Nuclear Extract at 3 dose levels on blood biomarkers | 25 weeks
  Serum Tau
To assess the impact of Thymus Nuclear Extract at 3 dose levels on blood biomarkers | 25 weeks
  Neurofilament Light
To assess the impact of Thymus Nuclear Extract at 3 dose levels on blood biomarkers | 25 weeks
  S100B
To assess the impact of Thymus Nuclear Extract at 3 dose levels on blood biomarkers | 25 weeks
  C-Reactive Protein
To assess the impact of Thymus Nuclear Extract at 3 dose levels on blood biomarkers | 25 weeks
  GFAP levels
To assess the impact of Thymus Nuclear Extract at 3 dose levels on blood biomarkers | 25 weeks
  Free and Total Triiodothyronine
To assess the impact of Thymus Nuclear Extract at 3 dose levels on blood biomarkers | 25 weeks
  Free and Total Thyroxine
To assess the impact of Thymus Nuclear Extract at 3 dose levels on blood biomarkers | 25 weeks
  Thyroid Stimulating Hormone
To assess the impact of Thymus Nuclear Extract at 3 dose levels on blood biomarkers | 25 weeks
  Triiodothyronine Uptake Test
To assess the safety and tolerability of Thymus Nuclear Extract at 3 dose levels | 25 weeks
  Gama-Glutamyl Transferase
To assess the safety and tolerability of Thymus Nuclear Extract at 3 dose levels | 25 weeks
  Uric Acid
To assess the impact of Thymus Nuclear Extract at 3 dose levels on blood biomarkers | 25 weeks
  Total Cortisol
To assess the impact of Thymus Nuclear Extract at 3 dose levels on blood biomarkers | 25 weeks
  C- Peptide
To assess the impact of Thymus Nuclear Extract at 3 dose levels on blood biomarkers | 25 weeks
  Lactate dehydrogenase
To assess the impact of Thymus Nuclear Extract at 3 dose levels on blood biomarkers | 12 weeks
  Corticoid-Binding Globulin
To assess the impact of Thymus Nuclear Extract at 3 dose levels on blood biomarkers | 12 weeks
  Free Cortisol Index

CONTACTS AND LOCATIONS:
Overall Officials: Bassem F. El-Khodor, PHD, Study Director — Standard Process Inc.
Locations (1):
- Model Research Center, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No